CLINICAL TRIAL: NCT02080507
Title: rTMS in Treatment Resistant Depression
Acronym: rTMSECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William McDonald MD, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00068138
Record Dates: First submitted 2014-03-04; First posted 2014-03-06 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Depression
Keywords: rTMS; depression; ECT
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Neuronetics rTMS stimulator (Active Comparator): Device: Active Neuronetics Transcranial Magnetic Stimulator. The Neuronetics transcranial magnetic stimulator is an FDA approved device. In the active group, magnetic power output will be delivered to the subject through the coils.
  Interventions: Device: Active Neuronetics rTMS stimulator
- Inactive Neuronetics rTMS stimulator (Sham Comparator): Device: Inactive Neuronetics Transcranial Magnetic Stimulator. The Neuronetics transcranial magnetic stimulator is an FDA approved device. In the inactive group, no magnetic power output will be delivered to the subject through the coils.
  Interventions: Device: Inactive Neuronetics rTMS stimulator

INTERVENTIONS:
Device: Active Neuronetics rTMS stimulator — In the active group, magnetic power output will be delivered to the subject through the coils.
  Other Names: Neuronetics
  Arms: Active Neuronetics rTMS stimulator
Device: Inactive Neuronetics rTMS stimulator — In the inactive group, no magnetic power output will be delivered to the subject through the coils.
  Other Names: Neuronetics
  Arms: Inactive Neuronetics rTMS stimulator

SUMMARY:
The purpose of this study is to determine the safety and efficacy of rTMS as an alternative treatment to ECT. The study will also provide data for a power analysis to support a larger clinical trial if there is evidence of a clinically relevant treatment effect.

DETAILED DESCRIPTION:
rTMS as an alternative to ECT

Background Electroconvulsive therapy (ECT) is highly effective in the treatment of severe depression (UK ECT Review Group, 2003). During the past decade, transcranial magnetic stimulation has emerged as a new anti-depressant treatment (e.g. Berman et al, 2000). Some randomized trials suggest that repetitive transcranial magnetic stimulation (rTMS) might be as effective as ECT in the treatment of non-psychotic depression (Grunhaus et al, 2000, 2003; Janicak et al, 2002; Rosa et all, 2003; Pridmore et al, 2000; Pridmore, 2000 ). Even at 3 and 6 month follow up, patients treated with rTMS continue to do as well as those treated with ECT (Dannon et al, 2002). A recent review also supported the efficacy of rTMS in treatment resistant depression (Lee et al, 2012). However, other reviews and meta-analyses show only moderate enthusiasm for transcranial magnetic stimulation as an alternative to ECT (e.g. Martin et al, 2003; Schlaepfer et al, 2003) and emphasize the need for further studies.

Given the small number of side effects and comparable efficacy to ECT, we would like to continue investigating rTMS as an alternative to ECT. The study will aim to compare the efficacy of sham vs. active rTMS in patients meeting standard criteria for ECT. In addition, the study will also determine the safety and efficacy of this trial and provide data for a power analysis to support a larger clinical trial if there is evidence of a clinically relevant treatment effect.

Our sample population will include 40 adult patients from the Emory University Outpatient Psychiatry Department and Atlanta community. Potential subjects may be identified by their treating physicians as potential subjects for the study and after obtaining permission from the patient, the physician will refer the patient to the research coordinator.

Subjects will enter a 4-week fixed-treatment phase and a variable 2-week extension for clinical improvers (defined below). Subject will receive rTMS treatment according the FDA approved protocol with treatments given five times a week daily Monday through Friday at 10 pulses/sec, 120% of motor threshold, and 3000 pulses/session for 4 weeks.

Patients who meet remission criteria (MADRS < 7 for one week, Riedel et al 2010) will be tapered from rTMS. Patients who do not show sufficient improvement at the end of the fixed 4-week period (defined as a < 30% drop from baseline in MADRS scores) will be discontinued. If patients improve sufficiently (i.e., > 30% reduction in MADRS score) but do not meet remission criteria, treatment will continue for up to 2 additional weeks (variable 2-week extension). In the variable phase, the MADRS assessments will be performed twice weekly and improvers, but nonremitters, will continue receiving treatment during the variable 2-week period if they show progressive improvement, defined as at least a 2-point MADRS score reduction at every other rating. The acute trial will be terminated when patients meet the stable remission criteria. The rTMS will then be tapered during a 3-week period.

Data Analysis Dichotomous outcomes (remission, response (defined as a 50% decrease in the baseline MADRS)) will be assessed using a logistic regression model (SAS Institute Inc., Cary, North Carolina) with independent variables of treatment (active vs. sham), medication resistance using the Antidepressant Treatment History Form (ATHF) (low vs. high), current depressive episode duration (log transformed) and age (continuous). The primary analysis will be conducted using the intention-to-treat (ITT) population, defined as all randomized patients who started at least 1 treatment session. All the statistical tests will be performed at the .05 significance level. Interactions were considered significant at the .15 significance level.

A primary purpose of the present study is to determine the safety and efficacy of this trial and provide data for a power analysis to support a larger clinical trial if there is evidence of a clinically relevant treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unipolar major depressive disorder or bipolar disorder, depressed phase and on medication to prevent a manic episode
* Pretreatment Montgomery Åsberg Depression Rating Scale (MADRS) score ≥ 20
* Over age 18 years
* Meeting criteria for ECT according to standards outlined in American Psychiatric Association Task Force on Electroconvulsive Therapy (2001) (American Psychiatric Association Task Force on Electroconvulsive Therapy: The Practice of Electroconvulsive Therapy: Recommendations for Treatment, Training and Privileging, Task Force Report on ECT, 2nd Edition. Washington, DC, American Psychiatric Association, 2001) and qualifying for ECT in the opinion of the study physician and the subject's psychiatric provider.
* Subjects may be on psychotropic medications including antidepressants, antipsychotics, benzodiazepines and anticonvulsants but the dosage of the medication must be stable for at least 6 weeks
* Able and willing to provide informed consent

Exclusion Criteria:

* Be pregnant or lactating, planning to become pregnant within the next three months or sexually active and not using birth control.
* 2. Diagnosis with the following conditions (current unless otherwise stated):

  1. Have a neurological disorder, including a history of seizures, cerebrovascular disease, primary or secondary tumors in central nervous system, stroke, cerebral aneurysm or movement disorder or any lifetime history of loss of consciousness due to head injury.
  2. Any current Axis 1 psychotic disorder (including substance-induced psychosis, psychotic disorder due to a medical condition, or major depression with psychotic features), as defined by the MINI ( Mini International Neuropsychiatric Interview; English Version 7.0.0 for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5); Copyright 1992---2014 Sheehan DV) at the screening visit;
  3. Any lifetime Axis 1 psychotic disorder (excluding substance-induced psychosis, or psychotic disorder due to a medical condition), or as defined by the MINI at the screening visit;
  4. Any current Axis II personality disorder that would interfere in the participation of the study as determined through medical history or in the opinion of the investigator;
  5. Have a current amnestic disorder, dementia, or delirium as defined by Montreal Cognitive Assessment of less than or equal to 16;
  6. Any illicit substance use as determined by positive toxicology screen for drugs of abuse; or alcohol and/or substance abuse or dependence within the past 3 months (90 days) as determined by the MINI at the screening visit
* Treatment histories including:

  1. Failure to clinically remit to an adequate trial of electroconvulsive therapy (ECT), defined as 8 bilateral or 10 unilateral treatments, in the current episode;
  2. Have failed prior treatment with vagal nerve stimulation (VNS);
  3. Prior treatment with TMS.
* Have active suicidal intent or plan as defined by a positive answer to questions 4 and/or 5 on the Columbia-Suicide Severity Rating Scale (CSSRS): Screening version; or more than one suicide attempt in lifetime; or a suicide attempt in the past twelve months; or in the Investigator's opinion, is likely to attempt suicide within the next six months.
* Participation in any drug or device clinical trial in the six weeks (42 days) prior to the screening visit and/or participation in another clinical trial for the duration of the study.
* Presence of any other condition or circumstance that, in the opinion of the investigator, has the potential to prevent study completion and/or to have a confounding effect on outcome assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William M McDonald, MD, Principal Investigator — Emory University
Locations (1):
- Emory University at Wesley Woods Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
We had not planned on sharing individual data with other researchers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited March 2014 through August 2015 from the Emory University Outpatient Psychiatry Department and the Atlanta community. Of the 16 participants who consented for participation, 12 began study treatment.
Pre-assignment Details: Participants taking psychotropic medications were required to be stable on a stable dose for at least six weeks.
Groups:
- Active Neuronetics rTMS Stimulator: Participants in this group were randomized to receive active repetitive transcranial magnetic stimulation (rTMS) five times a week at 10 pulses/sec, 120% of motor threshold, and 3000 pulses/session for 4 weeks.
- Inactive Neuronetics rTMS Stimulator: Participants in this group were randomized to receive sham repetitive transcranial magnetic stimulation (rTMS) five times a week at 10 pulses/sec, 120% of motor threshold, and 3000 pulses/session for 4 weeks.
Period: Overall Study
Arm/Group | Active Neuronetics rTMS Stimulator | Inactive Neuronetics rTMS Stimulator
Started | 5 | 7
Completed | 5 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Neuronetics rTMS Stimulator | Inactive Neuronetics rTMS Stimulator | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Depression Severity as Assessed by the Montgomery Åsberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. The MADRS-S instrument has nine questions, with an overall score ranging from 0 to 60 points. A higher score indicates greater depressive symptoms.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Neuronetics rTMS Stimulator | Inactive Neuronetics rTMS Stimulator
Number analyzed (Participants) | 5 | 7
units on a scale
  Baseline | 26.4 (3.14) | 29.29 (5.26)
  Week 6 | 11.5 (4.5) | 16.3 (4.03)

2. Secondary Outcome: Quality of Life Assessed by the Quality of Life Enjoyment and Satisfaction Questionnaire Short Form (Q-Les-SF) Score
Description: The Q-Les-SF assesses the degree of enjoyment and satisfaction experienced by individuals in various areas of daily functioning. The minimum raw score is 14, and the maximum score is 70. Higher scores indicate better satisfaction with life domains (physical health, feelings, work, household duties, school/course work, leisure time activities, and social relations).
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active Neuronetics rTMS Stimulator | Inactive Neuronetics rTMS Stimulator
Number analyzed (Participants) | 5 | 7
units on a scale
  Baseline | 37.14 (7.61) | 31.63 (15.41)
  Week 6 | 67.86 (7.14) | 40.18 (.89)

ADVERSE EVENTS:
Description: We used the clinicaltrials.gov definition for collection of adverse events
Arm/Group | Active Neuronetics rTMS Stimulator | Inactive Neuronetics rTMS Stimulator
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

LIMITATIONS AND CAVEATS:
The study sample was limited due to low recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes